CLINICAL TRIAL: NCT02290288
Title: Prospective Randomized Study for Vaginal Vault Prolapse After Hysterectomy: Comparison of a Vaginal and Laparoscopic Method With Validation of Translated Questionnaire for Symptoms and Quality of Life by Vaginal Prolapse.
Brief Title: Prospective Study for Vaginal Vault Prolapse After Hysterectomy: Comparison of Two Surgical Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Janusz Marcickiewicz, senior consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUREG-28601
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Vaginal Vault Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSF (Active Comparator): 1. vaginal surgery arm (SSF)
  Interventions: Procedure: vaginal surgery
- LSC (Active Comparator): laparoscopic surgery arm (LSC)
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: vaginal surgery
  Arms: SSF
Procedure: laparoscopic surgery
  Arms: LSC

SUMMARY:
The study is carried out at the Sahlgrenska University Hospital and the patient population consists of women referred with symptomatic and bothersome post-hysterectomy vaginal vault prolapse at least 1 cm above or beyond the hymeneal remnants. The interventions are either vaginal sacrospinousfixation or laparoscopic sacrocolpopexy following randomization to one of the types of surgery. The primary outcome is anatomical failure based on clinical assessment. Failure is defined clinically, according to the Pelvic Organ Prolapse Quantification system, as Ba, C or Bp at the hymen or below on maximum Valsalva maneuver one and two years after the surgery. Secondary outcomes are evaluation of continence, sexual function and prolapse symptoms based on validated questionnaires 1, 2, 5 and 10 years after the surgery.

DETAILED DESCRIPTION:
The lifetime risk for pelvic floor surgery for prolapse is likely to be between 10% and 15%, and a large number of patients who previously underwent hysterectomy develop vaginal vault prolapse. There is some evidence that about 2% of all women after hysterectomy would require a surgery for vault prolapse. There are many different techniques used for correction of vault prolapse but the evidence for them is lacking and the use is guided mainly by tradition at the singe institution.

There is some evidence indicating that laparoscopic surgery can be superior to the vaginal approach. Symptoms of prolapse are significantly associated with avulsion injury in patients after hysterectomy.

Our aim is to compare, with a 1- and 2-years follow-up examination in patients with post-hysterectomy prolapse, the efficacy of two standard surgical procedures for vaginal vault prolapse: sacrospinous vaginal colpopexy (the Richter procedure) with native tissue vaginal repair (sacrospinous fixation, SSF) and laparoscopic colposacropexy with mesh.

This is a single-center, randomized controlled trial of two standard surgical procedures for vaginal vault prolapse routinely used at our institution.Both procedures are designed to treat vault prolapse, one with mesh implantation through laparoscopy and the other with vaginal repairs and apical fixation to the sacrospinous ligament, usually on the right.

All patients referred to our gynecological unit (Ob/Gyn Department of Sahlgrenska University Hospital in Gothenburg) because of symptomatic vault prolapse and fulfilling the inclusions criteria are asked to participate in the study. Eligible for inclusion are: post-hysterectomy patients with at least two-compartment prolapse (with affected apical/vault compartment, stage II or higher on the Pelvic Organ Prolapse Quantification system (POP-Q)), suffering from symptoms of prolapse, requesting pelvic floor reconstructive surgery, and diagnosed with a vault prolapse. Excluded are: patients with prolapse and uterus in place, those not requesting pelvic floor surgery, patients who do not understand Swedish or are not capable to fulfill follow up procedure.

Patients undergo identical pre- and postoperative assessment procedures, including POP-Q examination on maximum Valsalva maneuver, which are archived on Case Report Form, and validated questionnaires PFDI-20, PFIQ-7 and PISQ-12. The study was approved by the regional ethics committee and all subjects obtain written informed consent to participate. To minimize the bias we decided that all the follow up examinations are going to be performed by the same gynecologist who do not perform the surgery.

All patients can end participation in the study at any moment.

The randomization process is carried out by computer, using patient social security number, at the time of enrollment (usually 2-3 months before the surgery). Patients are informed about their allocation after the randomization. Both procedures are performed by an experienced surgeon, with the patient under general anesthesia for the laparoscopic procedure and regional anesthesia for the sacrospinous fixation.

Patients are followed up at 3 months,1 year and 2 years postoperatively. These postoperative clinical examinations are performed by a single examiner, who had not been involved in the surgical procedures. The vaginal descent was assessed at maximum Valsalva maneuver.

In case of recurrence of prolapse and distressing symptoms which a patient desired to be resolved, a reoperation of prolapse is planned according to the clinical praxis at our department.

The primary outcome measure was anatomical failure based on clinical assessment. Failure was defined clinically as Ba, C or Bp at the hymen or below, on maximum Valsalva maneuver.

As secondary outcome measures we used a continence status, sexual function and prolapse symptoms based on validated questionnaires: Pelvic Floor Impact Questionnaire (PFIQ - 7), Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and quality of life based on Short Form (36) Health Survey.

The power calculation was based on the primary outcome measure and available data which led us to expect a failure rate of 25% in the sacrospinous fixation group and 10% failure in laparoscopy group. To detect an expected difference of 15% between the groups, with 80% power of the test 70 patients are required in each group.

ELIGIBILITY:
Inclusion Criteria:

* post-hysterectomy patients with at least two-compartment prolapse (with affected apical/vault compartment,
* stage II or higher on the Pelvic Organ Prolapse Quantification system (POP-Q)),
* suffering from symptoms of prolapse,
* requesting pelvic floor reconstructive surgery, and
* diagnosed with a vault prolapse.

Exclusion Criteria:

* patients with prolapse and uterus in place,
* those not requesting pelvic floor surgery,
* patients who do not understand Swedish or are not capable to fulfill follow up procedure

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
anatomical failure (Failure was defined clinically as Ba, C or Bp at the hymen or below, on maximum Valsalva maneuver.) | 1 year
  The primary outcome measure was anatomical failure based on clinical assessment. Failure was defined clinically as Ba, C or Bp at the hymen or below, on maximum Valsalva maneuver.

SECONDARY OUTCOMES:
continence status | 1 and 5 years
  continence status based on validated questionnaires: Pelvic Floor Impact Questionnaire (PFIQ - 7), Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
sexual function | 1 and 5 years
  sexual function based on validated questionnaires: Pelvic Floor Impact Questionnaire (PFIQ - 7), Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
prolapse symptoms | 1 and 5 years
  symptoms based on validated questionnaires: Pelvic Floor Impact Questionnaire (PFIQ - 7), Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12
quality of life | 1 and 5 years
  quality of life based on validated questionnaires: Pelvic Floor Impact Questionnaire (PFIQ - 7), Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and quality of life based on Short Form (36) Health Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Obst Gyn, Sahlgrenska University Hospital, Gothenburg, VGR, Sweden